CLINICAL TRIAL: NCT00460642
Title: Use of GnRH Antagonist (Cetrotide) Protocol, Instead of Agonist, to Prepare Recipients for Embryo Transfer
Brief Title: GnRH Antagonist to Prepare Recipients for Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Reproduction (IHR) (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IND 74,817
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Infertility
Keywords: Frozen embryo transfers (FET).; Egg donation (ED).; IVF.; ART.; Implantation.; GnRH antagonist.; Cetrotide.; Endometrial response.; Infertility treatments:; Transfer of embryos from egg donation (ED) to recipients.
MeSH Terms: conditions — Infertility | interventions — cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: GnRH Antagonist (Cetrotide)

SUMMARY:
26% of all ART cycles performed in the USA in 2003 (CDC data) are frozen embryo transfers (FET) and transfer of embryos resulting from egg donation (ED) to recipients. The typical protocol used to prepare a recipient for ET involves GnRH agonist (Lupron, Tap Pharmaceuticals) to down regulate the patient. A GnRH antagonist, such as Cetrotide (EMD Serono), is comparable to GnRH agonist and FDA approved to prevent spontaneous ovulation with ART treatment, and its usage decreases significantly the number of injections that the patient receives with treatment. The working hypothesis for this study is that the GnRH antagonist (Cetrotide) can be used instead of an agonist to achieve effective down regulation in FET and ED cycles. Presumably, patients will prefer Cetrotide over Lupron because of the markedly fewer injections required.

ELIGIBILITY:
Inclusion Criteria:

* History of infertility before cryopreserving the embryos or inability to conceive from her own oocytes (based on age and/or a serum FSH > 15 IU/L).
* Any patient desiring to become pregnant as a result of transferring frozen-thawed embryos generated using her own or donor oocytes.
* Subject is in good health as determined by the Investigator on the basis of medical history, physical examination and laboratory screening tests.
* A negative pregnancy test prior to starting treatment with estrogens.

Exclusion Criteria:

* Women with a history of liver and/or kidney disease
* Hypertension: systolic pressure over 180 mm Hg or diastolic pressure over 105 at any study visit, measured twice 6 hours apart despite active treatment for hypertension.
* Liver function tests of two times than the upper limit of normal
* Women with active sever endometriosis.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate

SECONDARY OUTCOMES:
Delivery Rate

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Tur-Kaspa, MD, Principal Investigator — President and Medical Director, Institute for Human Reproduction (IHR) and Director, Clinical IVF-PGD Program, Reproductive Genetics Institute (RGI).
Locations (2):
- United States (2):
  - Institute for Human Reproduction (IHR), Chicago, Illinois
  - Institute for Human Reproduction (IHR), Oakbrook Terrace, Illinois

REFERENCES:
- See also: Related Info — http://www.infertilityIHR.com